CLINICAL TRIAL: NCT05973175
Title: The RolE oF Androgen Excess in MUscle Energy MetaboLism in Women With PolyCystic Ovary Syndrome (The REFUEL PCOS) Study 1
Brief Title: REFUEL PCOS Study 1
Acronym: REFUEL-PCOS
Status: Recruiting | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University of Birmingham (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: REC 22/28
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Routine blood (cholesterol profile, HbA1C, LFTs, FBC, Renal profile) will be sent to the laboratory in the Beaumont Hospital for processing on the same day of sampling. Samples for steroid nontargeted metabolomics and muscle biopsy specimens will be stored in a -80C freezer in the research laboratory in the CRC building until analysis. Serum samples for targeted nontargeted metabolomics will be measured and analysed at the University of Birmingham by LC-MS/MS. Muscle biopsy specimens will undergo proteomic sequencing at the University College Dublin and metabolomic analysis at the University of Liverpool.
  The blood volume that will be collected is approximately 350ml. The amount collected for skeletal muscle tissue biopsies will be similar to half a grain of rice for each biopsies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with PCOS: The following inclusion criteria need to be met for the PCOS Study participants:
  * Women with a confirmed diagnosis polycystic ovary syndrome with androgen excess on clinical or biochemical grounds
  * BMI 20-40kg/m2
  * Age range 18-50 years
  * Ability to provide informed consent
- Women without PCOS (controls): The following inclusion criteria need to be met for the control Study participants:
  * No clinical features of possible polycystic ovary syndrome (absence of clinical features of androgen excess and ovulatory dysfunction).
  * BMI 20-40kg/m2
  * Age range 18-50 years
  * Ability to provide informed consent

SUMMARY:
Polycystic Ovary Syndrome (PCOS) affects 10% of all women, and it usually co-exists with high levels of male pattern hormones (also termed androgens). Women with PCOS are at increased risk of metabolic complications such as diabetes, non-alcoholic fatty liver disease, high blood pressure and heart disease. However, very little is understood about how androgen excess results in increased metabolic complications observed in women with PCOS.

The main aims of the REFUEL PCOS study are to compare markers of energy metabolism in women with PCOS to those without PCOS. This will allow the investigators to better understand metabolic risk by examining the relationship between androgen excess and energy metabolism. Skeletal muscle is an important site of energy metabolism, and emerging theories are that androgen excess impairs skeletal muscle energy balance and increases the risk of complications. Based on these emerging theories, the investigators want to investigate the effects of androgens on muscle energy metabolism. The investigators will also examine whether certain blood and urine result patterns can help identify differences in muscles energy metabolism and which women are at the highest risk of metabolic complications. This research will give insight into the metabolic risk associated with PCOS and treat and, where possible, prevent the development of metabolic disease in affected women.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a lifelong metabolic disorder, affecting 10-13% of all women, and is associated with a major healthcare and economic burden, estimated at $8 billion annually the US in 2020 (1, 2). Traditionally considered a reproductive disorder only, it is now increasingly clear that PCOS is associated with severe metabolic health consequences across the entire life course of women (3, 4). There is a two-fold increased risk of type 2 diabetes mellitus (T2DM) and nonalcoholic fatty liver disease, as well as emerging evidence of increased incidence of cardiovascular disease (CVD) (5-7). There are no disease-specific therapies to mitigate or treat metabolic risk in women with PCOS. This is consistently highlighted as the priority concern amongst PCOS patient advocacy groups.

Androgen excess is a cardinal feature of PCOS and circulating androgen burden is closely correlated with metabolic complications (5, 8-12). In women with PCOS, the risk of developing metabolic dysfunction is above that conferred by simple obesity, suggesting that androgen excess is a key player; however, a distinct mechanistic role for androgens in this process remains to be elucidated (13, 14). Androgen excess is associated with metabolically deleterious visceral fat accumulation and circulating testosterone levels correlate directly with the risk of T2DM and NAFLD. Muscle is a critical metabolic target tissue that plays a central role in energy metabolism through processes such as glucose uptake and oxidation, as well as oxidation of fatty acids to generate ATP in the mitochondria (15). Recent mechanistic data have shown that androgen excess is associated with changes in the transcriptional profile of skeletal muscle genes linked with metabolism and energy balance (15-17). Therefore, skeletal muscle is likely to represent an important site of crosstalk between androgen excess, disturbances in energy metabolism and risk of metabolic disease in PCOS.

Defective skeletal muscle glucose uptake is a key early step in the pathogenesis of insulin resistance in PCOS, and an early predictor of progression to overt type 2 diabetes mellitus. Impaired mitochondrial oxidation of free fatty acids in skeletal muscle, as well as other disturbances in skeletal muscle mitochondrial function such as oxidative phosphorylation, are increasingly implicated in the pathogenesis of metabolic disease such as T2DM (18-20). Abnormalities in skeletal muscle mitochondrial function have also been identified in small scale studies in women with PCOS, and were associated with impaired fatty acid oxidation, weight gain and an increased risk of diabetes (21, 22).

The investigators hypothesise that androgen-mediated disturbances in skeletal muscle energy balance play a major role in the pathogenesis of metabolic disease in women with PCOS. The investigators propose to test this using cross-sectional and interventional approaches utilising state-of-the-art metabolic phenotyping tools.

ELIGIBILITY:
Inclusion Criteria:

-

The following inclusion criteria need to be met for the PCOS Study participants:

* Women with a confirmed diagnosis polycystic ovary syndrome with androgen excess on clinical or biochemical grounds
* BMI 20-40kg/m2
* Age range 18-50 years
* Ability to provide informed consent

The following inclusion criteria need to be met for the control Study participants:

* No clinical features of possible polycystic ovary syndrome (absence of clinical features of androgen excess and ovulatory dysfunction).
* BMI 20.0-40kg/m2
* Age range 18-50 years
* Ability to provide informed consent

For participants with PCOS, a diagnosis of PCOS should be established on the basis of the Androgen Excess and PCOS (AE-PCOS) Society guidelines:

* Androgen excess (clinical and/or biochemical evidence)
* Chronic oligo-/anovulation (clinical and/or biochemical evidence)
* Clinical and/or biochemical exclusion of other conditions that could explain the above manifestation (e.g. congenital adrenal hyperplasia, Cushing's syndrome, Prolactinoma, adrenal and gonadal tumours)

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:

  * A confirmed diagnosis of diabetes
  * Current or recent (<3-months) use of weight loss medications
  * Current or recent use of oral contraceptive pill or hormone replacement therapy (within last 3-months)
  * Blood haemoglobin <11.0g/dL
  * History of alcoholism or a greater than recommended alcohol intake (recommendations > 21 units on average per week for men and > 14 units on average per week for women)
  * Haemorrhagic disorders
  * Treatment with anticoagulant agents
  * Other co-morbidities that in the view of the investigators may affect data collection
  * Any medical condition in the opinion of the investigator that might impact upon safety or validity of the results
  * Pregnancy or breastfeeding at the time of planned recruitment
  * A diagnosis of PCOS according to Rotterdam criteria where the patient does not have clinical or biochemical evidence of androgen excess
  * History of significant renal (eGFR<30) or hepatic impairment (AST or ALT >two-fold above ULN; pre-existing bilirubinaemia >1.2 ULN)
  * Any other significant disease or disorder that, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
  * Participants who have participated in another research study involving an investigational medicinal product in the 12 weeks preceding the planned recruitment
  * Glucocorticoid use via any route within the last six months
  * Current intake of drugs known to impact upon steroid or metabolic function or intake of such drugs during the six months preceding the planned recruitment
  * Use of oral or transdermal hormonal contraception in the three months preceding the planned recruitment
  * Use of contraceptive implants in the twelve months preceding the planned recruitment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Studying a female reproductive condition
Study Population: This study aims to recruit women with PCOS who have a BMI between 20 and 40kg/m2 with clinical or biochemical evidence of androgen excess. Their matched controls will have no clinical features of possible polycystic ovary syndrome (absence of clinical features of androgen excess and ovulatory dysfunction).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
To delineate the relationship between androgen excess and skeletal muscle energy metabolism in women | 2.5 years
  Baseline differences in the skeletal muscle proteome and differentially regulated pathways relating to mitochondrial function in hyperandrogenic women with PCOS compared to healthy controls

SECONDARY OUTCOMES:
Proteomic profiling of skeletal muscle biopsies will be integrated with serum steroid and non-targeted metabolome data to delineate the relationship between androgens and skeletal muscle energy metabolism in women | 2.5 years
  Differences in the non-targeted serum metabolome at baseline between women with PCOS and controls and Identification of differentially regulated pathways to facilitate targeted pathway analysis in future studies

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Collage Of Surgeons, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Clinical data (anthropomorphic and medical history) and data from in vivo phenotyping will be pseudonymised and uploaded to Redcap with biomaterial samples (urine, serum, muscle biopsy) stored in a bio-repository within the RCSI clinical research centre as per ethical approval. To ensure due process and aid sharing of the data the study will be registered online at (https://clinicaltrials.gov). Data will be shared upon request in keeping with Wellcome policy and as per REC guidance at the time of request post-publication of results.
Supporting Information: Study Protocol, SAP
Time Frame: 6 months following publication
Access Criteria: To ensure due process and aid sharing of the data the study will be registered online at (https://clinicaltrials.gov). Data will be shared upon request in keeping with Wellcome policy and as per REC guidance at the time of request post-publication of results.

REFERENCES:
- [Background] Riestenberg C, Jagasia A, Markovic D, Buyalos RP, Azziz R. Health Care-Related Economic Burden of Polycystic Ovary Syndrome in the United States: Pregnancy-Related and Long-Term Health Consequences. J Clin Endocrinol Metab. 2022 Jan 18;107(2):575-585. doi: 10.1210/clinem/dgab613. PMID 34546364
- [Background] Schiffer L, Arlt W, O'Reilly MW. Understanding the Role of Androgen Action in Female Adipose Tissue. Front Horm Res. 2019;53:33-49. doi: 10.1159/000494901. Epub 2019 Sep 9. PMID 31499495
- [Background] Nanba AT, Rege J, Ren J, Auchus RJ, Rainey WE, Turcu AF. 11-Oxygenated C19 Steroids Do Not Decline With Age in Women. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2615-2622. doi: 10.1210/jc.2018-02527. PMID 30753518
- [Background] Kumarendran B, O'Reilly MW, Manolopoulos KN, Toulis KA, Gokhale KM, Sitch AJ, Wijeyaratne CN, Coomarasamy A, Arlt W, Nirantharakumar K. Polycystic ovary syndrome, androgen excess, and the risk of nonalcoholic fatty liver disease in women: A longitudinal study based on a United Kingdom primary care database. PLoS Med. 2018 Mar 28;15(3):e1002542. doi: 10.1371/journal.pmed.1002542. eCollection 2018 Mar. PMID 29590099
- [Background] Legro RS, Arslanian SA, Ehrmann DA, Hoeger KM, Murad MH, Pasquali R, Welt CK; Endocrine Society. Diagnosis and treatment of polycystic ovary syndrome: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2013 Dec;98(12):4565-92. doi: 10.1210/jc.2013-2350. Epub 2013 Oct 22. PMID 24151290
- [Background] Randeva HS, Tan BK, Weickert MO, Lois K, Nestler JE, Sattar N, Lehnert H. Cardiometabolic aspects of the polycystic ovary syndrome. Endocr Rev. 2012 Oct;33(5):812-41. doi: 10.1210/er.2012-1003. Epub 2012 Jul 24. PMID 22829562
- [Background] Kempegowda P, Melson E, Manolopoulos KN, Arlt W, O'Reilly MW. Implicating androgen excess in propagating metabolic disease in polycystic ovary syndrome. Ther Adv Endocrinol Metab. 2020 Jun 24;11:2042018820934319. doi: 10.1177/2042018820934319. eCollection 2020. PMID 32637065
- [Background] Subramanian A, Anand A, Adderley NJ, Okoth K, Toulis KA, Gokhale K, Sainsbury C, O'Reilly MW, Arlt W, Nirantharakumar K. Increased COVID-19 infections in women with polycystic ovary syndrome: a population-based study. Eur J Endocrinol. 2021 May;184(5):637-645. doi: 10.1530/EJE-20-1163. PMID 33635829
- [Background] Barry JA, Kuczmierczyk AR, Hardiman PJ. Reporting the rates of depression in polycystic ovary syndrome (PCOS). J Sex Med. 2014 Jul;11(7):1882-3. doi: 10.1111/jsm.12503. Epub 2014 Mar 17. No abstract available. PMID 24636134
- [Background] Barry JA, Azizia MM, Hardiman PJ. Risk of endometrial, ovarian and breast cancer in women with polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod Update. 2014 Sep-Oct;20(5):748-58. doi: 10.1093/humupd/dmu012. Epub 2014 Mar 30. PMID 24688118
- [Background] O'Reilly MW, Kempegowda P, Jenkinson C, Taylor AE, Quanson JL, Storbeck KH, Arlt W. 11-Oxygenated C19 Steroids Are the Predominant Androgens in Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2017 Mar 1;102(3):840-848. doi: 10.1210/jc.2016-3285. PMID 27901631
- [Background] Escobar-Morreale HF, Alvarez-Blasco F, Botella-Carretero JI, Luque-Ramirez M. The striking similarities in the metabolic associations of female androgen excess and male androgen deficiency. Hum Reprod. 2014 Oct 10;29(10):2083-91. doi: 10.1093/humrep/deu198. Epub 2014 Aug 7. PMID 25104855
- [Background] O'Reilly MW, House PJ, Tomlinson JW. Understanding androgen action in adipose tissue. J Steroid Biochem Mol Biol. 2014 Sep;143:277-84. doi: 10.1016/j.jsbmb.2014.04.008. Epub 2014 Apr 28. PMID 24787657
- [Background] Nilsson E, Benrick A, Kokosar M, Krook A, Lindgren E, Kallman T, Martis MM, Hojlund K, Ling C, Stener-Victorin E. Transcriptional and Epigenetic Changes Influencing Skeletal Muscle Metabolism in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2018 Dec 1;103(12):4465-4477. doi: 10.1210/jc.2018-00935. PMID 30113663
- [Result] Skiba MA, Islam RM, Bell RJ, Davis SR. Understanding variation in prevalence estimates of polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod Update. 2018 Nov 1;24(6):694-709. doi: 10.1093/humupd/dmy022. PMID 30059968